CLINICAL TRIAL: NCT00518817
Title: The Cardiovascular Genetic and Therapeutic Implications of Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Baylor College of Medicine (Other)
Other Study IDs: Thrasher
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Muscular Dystrophy; Dilated Cardiomyopathy; Heart Failure
Keywords: Dystrophy; Cardiomyopathy
MeSH Terms: conditions — Muscular Dystrophies; Cardiomyopathy, Dilated; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will have significant impact on muscular dystrophy patients as it promotes early screening for heart disease. With early identification, beneficial medical therapy can be started sooner, resulting in restoring and maintaining normal heart function. This is critical to the survival of these patients. We have reported previously that heart failure in all patients may have common mechanisms, the "final common pathway". Heart failure is a significant health problem with 5 million people in the US carrying the diagnosis and accounting for 12-15 million office visits and 6.5 million hospital days per year. The number of deaths from heart failure continues to increase. The data from this study could impact patients worldwide with heart failure by offering new insight into an ever-growing disease population and lead to significant changes in how they are currently treated.

DETAILED DESCRIPTION:
Objective(s) and Hypothesis(es): The objectives to be evaluated are as follows:

Specific Hypothesis #1: Heart disease, specifically dilated cardiomyopathy, can be identified early in patients with muscular dystrophy and allow for earlier institution of medical therapies

Specific Hypothesis #2: Non-invasive testing via magnetic resonance imaging (MRI) and echocardiography can identify early systolic and diastolic dysfunction in patients with muscular dystrophy as well as document structural changes ("Reverse remodeling") following institution of medical therapy

Specific Hypothesis #3: Serologic testing can identify early cardiac dysfunction prior to changes on magnetic resonance imaging or echocardiogram that can predict disease onset, risk stratify future cardiac morbidity and mortality, and response to medical therapy

Specific Hypothesis #4: Specific dystrophin mutations can be identified that predict the onset or protection against dilated cardiomyopathy

Specific Hypothesis #5: Construction and maintenance of a database of patients with muscular dystrophy can be established that will allow for future research in patients with muscular dystrophy, specifically in the area of gene therapy

Specific Hypothesis #6: Quality of life in patients with cardiac disease can be assessed and used to modulate therapy and also allow for noncardiac directed therapies that will improve overall well-being

Specific Hypothesis #7: Further understanding of neurohormonal profiles, responses to medical therapy, and dystrophin mediated cardiomyopathy will impact all patients with heart failure world-wide

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of muscular dystrophy.

Exclusion Criteria:

* Patients that do not carry the diagnosis of muscular dystrophy.

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John L Jefferies, MD, Principal Investigator — Baylor College of Medicine; Jeffrey A Towbin, MD, Study Director — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States